CLINICAL TRIAL: NCT03757910
Title: Amyloid Brain Positron Emission Tomography (PET) Imaging With 11C-PIB and Tau PET Imaging With 18F-MK-6240 in the Diabetes Prevention Program Outcomes Study.
Brief Title: Brain Imaging in the Diabetes Prevention Program Outcomes Study
Acronym: DPPOS-Brain
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Difficulty recruiting due to the COVID-19 pandemic and end of funding
Sponsor: José A. Luchsinger (Other)
Collaborators: Albert Einstein College of Medicine (Other); George Washington University (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor-Investigator, José A. Luchsinger, Professor of Medicine and Epidemiology, Columbia University
Organization: Columbia University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: AAAS1176; 3U01DK048404-25S1 (NIH)
Record Dates: First submitted 2018-11-27; First posted 2018-11-29 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-03

CONDITIONS: Alzheimer Disease
Keywords: Metformin; Pre-diabetes; Type 2 diabetes; DPPOS
MeSH Terms: conditions — Alzheimer Disease; Glucose Intolerance; Diabetes Mellitus, Type 2 | interventions — 2-(4'-(methylamino)phenyl)-6-hydroxybenzothiazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- DPPOS Exposed to Metformin (Experimental): DPPOS participants with exposure to metformin will be scanned with 18F-MK-6240 and 11C-PIB.
  Interventions: Drug: 18F-MK-6240; Drug: 11C-PIB
- DPPOS Exposed to Placebo (Active Comparator): DPPOS participants with no exposure to metformin but only placebo will be scanned with 18F-MK-6240 and 11C-PIB.
  Interventions: Drug: 18F-MK-6240; Drug: 11C-PIB

INTERVENTIONS:
Drug: 18F-MK-6240 — This radiotracer will be used to detect Tau.The injected activity will equal 5 millicuries (mCi).
Drug: 11C-PIB — This radiotracer will be used to detect amyloid. Participants will be injected with an intravenous bolus of up to 5-15 mCi.
  Other Names: 11C-Pittsburgh Compound B

SUMMARY:
This is a cross-sectional pilot study of Alzheimer's disease (AD) brain imaging biomarkers in Diabetes Prevention Program (DPP) outcomes study (DPPOS) participants from the New York City sites (Columbia and Einstein), comparing 10 persons originally randomized to metformin and 10 persons randomized to placebo in DPP. All study procedures will be conducted at Columbia University Irving Medical Center. Eligible participants will receive a PET scans and a brain MRI, which may be conducted in one, two, or three separate visits.

DETAILED DESCRIPTION:
Hyperinsulinemia is believed to increase the risk of Alzheimer's dementia through both cerebrovascular and A related mechanisms, and this hypothesis has prompted testing strategies related to hyperinsulinemia and diabetes in the prevention and treatment of Alzheimer's dementia.These strategies usually entail improving insulin sensitivity to lower insulin and glucose levels, such as lifestyle (diet and exercise) and metformin, which were effective strategies for preventing diabetes in the DPPOS. There are conflicting data relating metformin with increased AD risk, and this needs to be clarified in DPPOS. Several laboratory and human studies have suggested that metformin increases the risk of Alzheimer's dementia, but this is countered by other studies indicating that it is beneficial. Preliminary data in humans and animals support the beneficial effects of metformin on Alzheimer's dementia risk.

ELIGIBILITY:
Inclusion Criteria:

* Active participants in the Diabetes Prevention Program Outcomes Study (DPPOS) in New York City originally randomized to metformin or placebo
* 60 years and older

Exclusion Criteria:

* Known dementia
* Contraindications to magnetic resonance imaging (MRI)
* Contraindications to radio-contrast agents.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Brain Amyloid SUVR | Up to 1 hour post-injection
  Whole brain amyloid (11C-PIB) standardized uptake volume ratio (SUVR)
Brain Tau SUVR | Up to 1 hour post-injection
  Tau (18F-MK-6240) SUVR in medial and inferior temporal lobes

SECONDARY OUTCOMES:
Hippocampal Cortical Thickness | Up to 1 hour post-injection
  Thickness in the hippocampal cortex
White Matter Hyper Intensity Volume | Up to 1 hour post-injection
  Volume of brain white matter hyper-intensities

CONTACTS AND LOCATIONS:
Overall Officials: Jose A. Luchsinger, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided